CLINICAL TRIAL: NCT07382336
Title: A Mobile Application for Early Detection and Symptoms Trajectories of Postpartum Depression Using Ecological Momentary Assessment (EMA): A Prospective Cohort Validation Study
Brief Title: A Mobile Application for Early Detection and Symptoms Trajectories of Postpartum Depression Using Ecological Momentary Assessment (EMA)
Acronym: EMA For PND
Status: Recruiting | Type: Observational
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, LIN Jingxia Jessie, Assistant Professor, The Hong Kong Polytechnic University
Other Study IDs: 20211291; 20211291 (Other Grant/Funding Number: Hong Kong Health and Medical Research Fund)
Record Dates: First submitted 2026-01-25; First posted 2026-02-02 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Postpartum Depression (PPD)
Keywords: Ecological momentary assessment; Postpartum depression
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ecological momentary assessment group
  Interventions: Diagnostic Test: Ecological momentary assessment and retrospective assessment

INTERVENTIONS:
Diagnostic Test: Ecological momentary assessment and retrospective assessment — The intervention includes daily EMA components, and monthly retrospective assessments.

SUMMARY:
This pilot study will recruit 120 perinatal pregnant women and follow them up for 6 months. Both momentary and retrospective assessments of emotional well-being and psychosocial factors will be conducted on a mobile application. We aim to understand the symptom trajectories and provide evidence for effective individualized interventions.

DETAILED DESCRIPTION:
The proposed study addresses the knowledge gaps regarding the validity of mobile-based ecological momentary assessment (EMA) for dynamic patterns of mood symptoms and associated factors in women during pregnancy through postnatal period. The investigators hypothesize that the validity of mobile-based EMA is appropriate in women during pregnancy through postnatal period and that participants will exhibit at least two trajectories of depressive symptoms with high and low severity over a six-month period from the third trimester to three months postpartum. This prospective study using single group design will recruit 120 pregnant women for a six-month period. Clinical and self-rating assessments of mood symptoms and lifestyle information will be conducted on a mobile application. There will be a total of six periods EMA assessments and seven retrospective assessments. Six EMA questions for mood, sleep, exercise, physical well-being, and environmental context will be administered three times daily for five consecutive days, and the Edinburgh Postnatal depression Scale will be assessed at baseline and each month during the six-month period. Descriptive and inferential statistics will be used to examine the feasibility and validity of mobile-based EMA. Hierarchical cluster analysis and multiple regression model will be used to identify trajectories of depressive symptoms, and associated factors.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in their first and second trimesters.
* Aged 18 years and older.
* Able to read and understand Chinese
* Own a smartphone with iOS or Android system.

Exclusion Criteria:

* Psychiatric diagnosis (e.g., schizophrenia, intellectual disability or mood disorders), comorbid brain conditions (history of epilepsy, stroke, or brain tumors), or learning disabilities.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Females
Study Population: Perinatal women
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Ecological Momentary Questions (Mood) | Three momentary assessments per day for five days in each month for 6 months, displayed randomly within each of the following intervals: 0900-1300, 1300-1800 and 1800-0000.
  Three momentary questions will be administered to assess participants' mood-two yes/no Whooley questions for depression, one question about anxiety, which questions will be mapped onto a five-point pictorial scale, ranging from 1 (lowest) to 5 (highest) points. The higher score means worse outcome.
Edinburgh Postnatal Depression Scale (EPDS) | At the baseline and the end of each of the 6 months in the period.
  Measures postnatal depression. Each item scores 0-3, and the total score ranges from 0 (min) to 30 (max). Higher score means worse depressive symptoms.

SECONDARY OUTCOMES:
Ecological Momentary Questions (Lifestyle and Physical Wellbeing) | Three momentary assessments per day for five days in each month for 6 months, displayed randomly within each of the following intervals: 0900-1300, 1300-1800 and 1800-0000.
  Three momentary questions will be administered to assess participants' sleep, exercise and physical pain/fatigue; they will be either mapped onto a five-point pictorial scale, ranging from 1 (min) to 5 (max) points (sleep) or presented using yes/no questions (exercise and physical pain/fatigue). For sleep, the higher score means better outcome.
Ecological Momentary Questions (Contextual) | Three momentary assessments per day for five days in each month for 6 months, displayed randomly within each of the following intervals: 0900-1300, 1300-1800 and 1800-0000.
  Two contextual questions will be administered to complement the momentary mood questions. They will assess participants' location and the activity in which they are engaged at the time they answer the six momentary questions.
Depression Anxiety and Stress Scale 21 (DASS-21) | At the baseline and the end of each of the 6 months in the period
  Measures stress symptoms. Each item scores 0-3, the total score for stress ranges from 0 (min) to 21 (max). Higher score means worse symptoms of stress.
Post-study acceptance survey | The survey will be conducted via online when the participants complete 6-month study.
  A questionniare at the end of the six-month study period to assess the acceptability of the app to participants in the context of their prenatal and postnatal care and to collect feedback about their experience with the app.

CONTACTS AND LOCATIONS:
Overall Officials: Jessie LIN, PhD, Study Chair — Department of Rehabilitation Sciences, The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
May need to seek approval of the funding body.